CLINICAL TRIAL: NCT02175537
Title: Microclinic Social Induction Pilot Intervention for Diabetes and Obesity Management in Qatar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Microclinic International (Other)
Collaborators: Qatar University (Other); Qatar Foundation (Unknown); Qatar Diabetes Association (Unknown); Qatar Supreme Council of Health (Unknown); Harvard School of Public Health (HSPH) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NPRP2014-2017
Record Dates: First submitted 2014-06-18; First posted 2014-06-26 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes Mellitus, Type II; Overweight and Obesity; Hypertension; Behavioral Lifestyle Change; Social Change
Keywords: Diabetes Mellitus, Type II; Disease management; Obesity; Social Network; Chronic disease; Prevention and control; Education
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity; Hypertension; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Microclinic social induction training (Experimental): BMI of 30 and over; or BMI of 25 and over and self-reported pre-diabetes or type II diabetes will receive the Microclinic Social Induction Diabetes and Obesity Program. The intervention is a training on diabetes self-management, disease monitoring, diabetes prevention, prevention of complications, health behavior change, and social network supports in order to improve chronic disease risk factors.
  Interventions: Behavioral: Microclinic Social Induction Diabetes and Obesity Program
- Controls (No Intervention): Receiving no intervention but parallel primary and secondary outcome measures as intervention study arm

INTERVENTIONS:
Behavioral: Microclinic Social Induction Diabetes and Obesity Program — Microclinics consist of 2-8 individuals from pre-existing social networks (friends, relatives, coworkers, neighbors, etc) that voluntarily participate in ongoing education and medical monitoring from local health care professionals, learning and practicing diabetes management strategies, sharing much-needed medical supplies, and exchanging social support.
  Arms: Microclinic social induction training

SUMMARY:
The purpose of the study is to pilot-phase test the effectiveness of the microclinic social induction model and its effects on behavioral and metabolic outcomes in different levels of social and familial relationships in Qatar. The investigators novel microclinic model is based on the principle that both healthy and unhealthy behaviors spread through preexisting social networks. A microclinic is a small group of approximately 2-8 friends or family members who are taught to modify their own behaviors as well as the behaviors of those around them, with a particular focus on the four "M's": Meals, Movement, Monitoring, and Medication. More than social support groups or peer-to-peer interventions, the microclinic model is unique in its focus on the long-term propagation of healthy behaviors throughout a participant's entire social network. Qatar is uniquely positioned (with its central geographic location in the Gulf region and its leadership in science and education) to spearhead a regional intervention focused on managing and preventing diabetes in the Gulf region.

DETAILED DESCRIPTION:
This pilot study, "Microclinic Social Induction Intervention for Diabetes and Obesity Management in Qatar," is a two-arm randomized controlled trial of a 7-week condensed intervention to evaluate the efficacy of the microclinic social induction model on propagating lifestyle changes and in improving glycemic and metabolic control in Doha, Qatar.

The microclinic social induction model leverages different levels of social and familial relationships to positively influence behaviors relating to diabetes and other metabolic conditions through small treatment units called 'microclinic groups,' consisting of 2-8 peers and family members of the same social network. The intervention model brings microclinic groups to a larger classroom network (~25 people/class) where each class shares access to a culturally salient diabetes educational curriculum and group support to promote health behavior changes such as improvement in diet, exercise, medication adherence, and blood pressure management to then influence better glycemic and metabolic control.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Mentally competent
* Body Mass Index of 30 or higher
* Body Mass Index of 25 or higher and self-reported pre-diabetes or type II diabetes

Exclusion Criteria:

* They do not meet the above criteria
* They are pregnant
* They have significant medical complications that prevent them from making changes to diet or level of physical activity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Weight | Weekly measurements between baseline and end of trial after 7 weeks
  Change in body weight (and BMI)
HbA1c | Baseline, end of trial after 7 weeks
  Change in HbA1c from baseline to end of 7-week pilot phase.
Waist circumference | Baseline, 4th-week midpoint, 7th-week final

SECONDARY OUTCOMES:
Blood Pressure | Baseline, 4th-week midpoint, 7th-week final
  Systolic and diastolic blood pressure changes
Health Profile Survey | Baseline, end of trial after 7 weeks.
  Change in overall health seeking and health maintenance behaviors.

OTHER OUTCOMES:
Social Network Relationships | Baseline, end of trial after 7 weeks.
  Changes in degree of interpersonal health support relationships as assess on Social Network Matrix instrument

CONTACTS AND LOCATIONS:
Overall Officials: Eric L Ding, PhD, Principal Investigator — Harvard School of Public Health (HSPH); Daniel Zoughbie, DPhil, Principal Investigator — Microclinic International
Locations (1):
- Qatar Diabetes Association, Doha, Qatar

REFERENCES:
- See also: Related info on Microclinic International — http://www.microclinics.org/